CLINICAL TRIAL: NCT06118710
Title: Evaluation of the Omission of Dexamethasone in Premedication Regimens During Paclitaxel Treatment
Acronym: DEXASTOP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Roelof W.F. van Leeuwen, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU_CT 2023-507481-43-00
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Dexamethasone; Histamine H1 Antagonists

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, randomized, non-inferiority trial.
Masking Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental premedication regimen (Experimental): Local standard of care premedication regimen with an Histamine-1 antagonist (e.g. clemastine or cetirizine) without dexamethasone
  Interventions: Drug: H1 Antihistaminics
- Local standard of care premedication regimen (Active Comparator): Local standard of care premedication regimen with an Histamine-1 antagonist (e.g. clemastine or cetirizine) with dexamethasone
  Interventions: Drug: Dexamethasone; Drug: H1 Antihistaminics

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone prior to paclitaxel infusion according to local care standards.
  Arms: Local standard of care premedication regimen
Drug: H1 Antihistaminics — Clemastine or Cetirizine prior to paclitaxel infusion according to local care standards

SUMMARY:
This prospective multicenter randomized non-inferiority trial aims to assess whether omitting dexamethasone from the premedication regimen during paclitaxel-based chemotherapy is non-inferior to the standard of care regimen that includes dexamethasone, based on the incidence of clinically relevant hypersensitivity reactions (HSRs) of grade ≥3 as per CTCAE v5.0. With a study population of 500 adult patients with solid tumors, the trial will also investigate secondary endpoints including the severity and incidence of HSRs of any grade, the number of paclitaxel administrations until the first HSR, the impact on patients' quality of life, adverse events related to dexamethasone, and the cost-effectiveness of the two premedication regimens from healthcare and societal perspectives.

DETAILED DESCRIPTION:
Rationale Dexamethasone is administered alongside a H1-antagonist (e.g. cetirizine) to prevent hypersensitivity reactions (HSRs) during paclitaxel chemotherapy. However, the rationale seems limited and several studies have demonstrated no increase in HRSs after discontinuation of dexamethasone after the second paclitaxel administration. In addition, two studies have demonstrated the feasibility of lower doses of dexamethasone in paclitaxel premedication regimens. Furthermore, there seems to be no statistically significant association between the administration route (Intravenous (IV) or oral) or dose of dexamethasone and the HSR rate.

Dexamethasone may lead to serious side effects such as hyperglycemia, immune suppression, mood disturbances, sleeping disorders, and weight gain, thereby negatively affecting the patient's health-related quality of life (HRQoL).

Discontinuing dexamethasone might result in improved HRQoL, decreased healthcare costs, and more efficient premedication regimens. However, no head-to-head studies on dexamethasone's added value in preventing paclitaxel-induced HSRs have been performed. Therefore, the aim of our study is to demonstrate that the premedication regimen without dexamethasone is non-inferior to the standard of care premedication regimen with dexamethasone, based on the incidence of paclitaxel-induced HSRs (Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade ≥3).

Objective The primary objective is to evaluate the incidence of clinically relevant HSRs (grade ≥3 as per Common Terminology Criteria for Adverse Events; CTCAE version 5.0) during paclitaxel-based chemotherapy with a standard of care premedication regimen with dexamethasone compared to an experimental premedication regimen without dexamethasone.

Secondary objectives are: To determine the incidence and severity of HSRs (any grade) during paclitaxel-based chemotherapy with a standard of care premedication regimen with dexamethasone compared to an experimental premedication regimen without dexamethasone; To determine the number of paclitaxel administrations and cumulative dose until the first HSR occurrence (any grade); To determine the effect of dexamethasone omission on the patient's quality of life; To determine the incidence and severity of adverse events related to dexamethasone; To determine the cost-effectiveness of the premedication regimens with and without dexamethasone from a healthcare and societal perspective.

Main trial endpoints The primary outcome will be the percentage of patients who experience a clinically relevant HSR (CTCAE grade ≥3) during paclitaxel infusion (Yes/No), determined prospectively by the oncology medical staff (e.g. oncologist).

Secondary trial endpoints Secondary outcomes are: The severity of the HSR grades as defined by (CTCAE v.5.0); The incidence of the HSRs (all grades) as defined by (CTCAE v.5.0); The percentage (%) of patients that can be rechallenged (conform standard of care) after the occurrence of an HSR with or without dexamethasone; The number of paclitaxel administrations and cumulative dose (mg) until the first HSR occurrence; The incidence and severity of adverse events related to dexamethasone measured through the validated Dexamethasone Symptom Questionnaire (DSQ)(21); The patient quality of life measured using the EuroQol-5 dimensions-5 levels (EQ-5D-5L) and European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C-30) scorings tools); The costs of the paclitaxel premedication regimen with and without dexamethasone from a healthcare and societal perspective.

Trial design This is a prospective, multicenter, randomized, non-inferiority trial.

Trial population In total, 500 patients (≥18 yo) with solid tumors (any indication) for whom paclitaxel-based chemotherapy is considered standard treatment will be included.

Interventions Eligible patients will be randomized 1:1 to receive either the local standard of care premedication regimen with dexamethasone or the experimental premedication regimen without dexamethasone during five administrations of paclitaxel. Patients will start with paclitaxel treatment on the physicians recommended dose as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosis of a solid tumor with planned treatment with paclitaxel-based chemotherapy for any indication and with any dose.
* Mastery of Dutch language
* Able and willing to give written informed consent.

Exclusion Criteria:

* Prior treatment with a paclitaxel-based regimen;
* An indication for paclitaxel in combination with moderately or highly emetogenic chemotherapy that mandates the use of dexamethasone as an anti-emetic medication (e.g., carboplatin AUC>4);
* Known hypersensitivity to paclitaxel, carboplatin, cetirizine, granisetron, ondansetron or excipients (e.g., benzyl alcohol);
* Concomitant use of any systemic corticosteroid for any indication other than paclitaxel premedication;
* Women with confirmed and ongoing pregnancy;
* Already participating in an exercise trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the percentage of patients who experience a clinically relevant HSR (CTCAE grade ≥3) during paclitaxel infusion (Yes/No), determined prospectively by the oncology medical staff (e.g. oncologist). | Throughout the entire duration of the study, spanning five cycles of paclitaxel treatment
  The primary outcome is the percentage of patients who experience a clinically relevant HSR (CTCAE grade ≥3) during paclitaxel infusion (Yes/No), determined prospectively by the oncology medical staff (e.g. oncologist).

SECONDARY OUTCOMES:
The severity of the HSR grades as defined by (CTCAE v.5.0); | Throughout the entire duration of the study, spanning five cycles (each cycle is 7 days) of paclitaxel treatment
  The severity of the HSR grades as defined by (CTCAE v.5.0);
The incidence of the HSRs (all grades) as defined by (CTCAE v.5.0); | Throughout the entire duration of the study, spanning five cycles (each cycle is 7 days) of paclitaxel treatment
  The incidence of the HSRs (all grades) as defined by (CTCAE v.5.0);
The percentage (%) of patients that can be rechallenged (according to standard of care procedures) after the occurrence of an HSR with or without dexamethasone; | Throughout the entire duration of the study, spanning five cycles (each cycle is 7 days) of paclitaxel treatment
  The percentage (%) of patients that can be rechallenged (according to standard of care procedures) after the occurrence of an HSR with or without dexamethasone;
The incidence and severity of adverse events related to dexamethasone measured through the validated Dexamethasone Symptom Questionnaire (DSQ) | Throughout the entire duration of the study, spanning five cycles (each cycle is 7 days) of paclitaxel treatment
  The incidence and severity of adverse events related to dexamethasone measured through the validated Dexamethasone Symptom Questionnaire (DSQ)
The patient quality of life measured using the EuroQol-5 dimensions-5 levels (EQ-5D-5L) scorings tools. | Throughout the entire duration of the study, spanning five cycles (each cycle is 7 days) of paclitaxel treatment
  The patient quality of life measured using the EuroQol-5 dimensions-5 levels (EQ-5D-5L) and European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C-30) scorings tools)
The patient quality of life measured using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C-30) scorings tools. | Throughout the entire duration of the study, spanning five cycles (each cycle is 7 days) of paclitaxel treatment
  The patient quality of life measured using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C-30) scorings tools.
• The total cost of treatment of both premedication regimens from a healthcare and societal perspective. | Throughout the entire duration of the study, spanning five cycles (each cycle is 7 days) of paclitaxel treatment
  • The total cost of treatment of both premedication regimens from a healthcare and societal perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zietse M, Aalders LC, Spierings LEAMM, De Rouw N, Dercksen W, Dalm VASH, Oomen-de Hoop E, Thielen FW, Koch BCP, Mathijssen RHJ, van Doorn L, Leeuwen RWFV. Omission of dexamethasone in paclitaxel premedication regimens: protocol of the multicentre, randomised, non-inferiority DEXASTOP trial. BMJ Open. 2025 Apr 25;15(4):e102770. doi: 10.1136/bmjopen-2025-102770. PMID 40280620